CLINICAL TRIAL: NCT02128633
Title: EFFECTIVENESS OF A HOMECARE DESENSITIZER FOR PATIENTS WITH DENTIN HYPERSENSITIVITY
Brief Title: Effectiveness of a Homecare Dentin Hypersensitivity Gel
Acronym: ECR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Franciscan University Center (Other)
Responsible Party: Principal Investigator, Fabricio Batistin Zanatta, Orientador principal, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM_DH_2014
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Dentin Sensitivity
Keywords: Dentin hypersensitivity; Dentin Sensitivities
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride; Oxalic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): Individuals that were randomized for treatment " A " . The product tested were always delivered in a transparent plastic syringe with 10 mls marking identified by the letters " A " . The syringes were given to individuals in an opaque plastic envelope sealed and delivered along with a reminder of the correct way to use the products. Guidance for the use of substances was to make application with a new toothbrush, 1 time a day (at night, before bed, after brushing the teeth) with the product received, for 1 minute and the amount of 0.25 g (0.5 ml) of the product as the demarcation the syringe. It was recommended that after using the products, they were expelled without rinsing the oral cavity with water (Placebo gel).
  Interventions: Drug: placebo gel
- Experimental gel (Experimental): Individuals that were randomized for treatment " B " - The product was delivered in a transparent plastic syringe with 10 mls identified by the letter " B ". The syringes were given to individuals in an opaque plastic envelope sealed and with a reminder of the correct way to use the products. Guidance for the use of substances was to make application with a new toothbrush, 1 time a day (at night, before bed, after brushing the teeth) with the product received, for 1 minute and the amount of 0.25 g (0.5 ml) of the product as the demarcation the syringe. It was recommended that after using the products, they were expelled without rinsing the oral cavity with water (5% sodium fluoride, potassium oxalate 5%, strontium chloride 10% ) .
  Interventions: Drug: 5% sodium fluoride, potassium oxalate 5%, strontium chloride 10%
- Positive control (Active Comparator): Individuals that were randomized for treatment " C " . The product tested were always delivered in a transparent plastic syringe with 10 mls marking identified by the letters " C " . The syringes were given to individuals in an opaque plastic envelope sealed and delivered along with a reminder of the correct way to use the products. Guidance for the use of substances was to make application with a new toothbrush, 1 time a day (at night, before bed, after brushing the teeth) with the product received, for 1 minute and the amount of 0.25 g (0.5 ml) of the product as the demarcation the syringe. It was recommended that after using the products, they were expelled without rinsing the oral cavity with water (Fluoride neutral NaF gel 2 %).
  Interventions: Drug: Fluoride neutral NaF gel 2 %

INTERVENTIONS:
Drug: placebo gel — Manipulated at Novaderme ®, Santa Maria, RS, Brazil.
  Other Names: The product (Treatment "A") was manipulated.
  Arms: placebo
Drug: 5% sodium fluoride, potassium oxalate 5%, strontium chloride 10% — Manipulated at Novaderme ®, Santa Maria, RS, Brazil.
  Other Names: The product (Treatment "B") was manipulated with the three active agents.
  Arms: Experimental gel
Drug: Fluoride neutral NaF gel 2 % — The product had similar appearance and viscosity than others.
  Other Names: Flugel®, DFL, Rio de Janeiro, Brazil;
  Arms: Positive control

SUMMARY:
Aim: To evaluate the effectiveness of a desensitizing gel for topical and home use in the treatment of dentin hypersensitivity (DH) through a randomized clinical trial, double-blind, with three parallel treatment. Methods: 126 subjects were divided into three groups: placebo gel (PG), test gel (TG) (5% sodium fluoride, potassium oxalate 5%, strontium chloride 10%) and sodium fluoride gel (2% FG ). The measurement of DH was performed by a single examiner blinded by the visual analog scale (VAS) after tactile, thermal and osmotic stimuli in the Baseline, 7, 15 and 30 days.

DETAILED DESCRIPTION:
STUDY POPULATION

The sample was recruited in clinics of the School of Dentistry at the Franciscan University Center and the specialization course in Periodontics at the University of Inga - . St. Mary (UNINGÁ). After the selection of patients, issues related to medical and dental history were collected through a semi-structured questionnaire. Subsequently, in teeth included in the study, conducted the assessment of gingival recession and the width and depth (in the case of the presence of non-carious cervical lesions) in millimeters with a millimeter probe type Willians (Neumar®, São Paulo , SP , Brazil) to estimate the area of wear in mm3. Still, the recession of each subject was classified according to its probable etiology and associated with periodontal disease (recession on the buccal surface and proximal surfaces on the teeth with DH in a subject with attachment loss ≥ 3 mm and probing depth ≥ 3mm affecting interproximal sites of two non-adjacent or more teeth). The others were considered associated with brushing trauma.

SAMPLE SIZE

The calculation of sample size was based on a clinically significant difference between two groups in the reduction of DH after stimulation with compressed air (mean difference of 20 mm and a standard deviation of 30mm on a visual analog scale). Considering a significance level of 5%, power 80% of the study and design in parallel, were estimated at least 36 patients for each group. Considering a dropout rate of 15% of the study, the size was increased to 42 eligible individuals per group.

RANDOMIZATION

Eligible patients were randomized in blocks in the form of allotment into three groups. For this, they were placed in a manila envelope with 2 papers with each letter "A", "B" and "C". The draw was always held by a third person (R.A.), which also gave the gel to the patient. All envelopes were sequentially numbered and were sealed. The sequential envelope was opened only after the draw of the six letters of the previous envelope.

BLINDING

The study was completely double-blind. At no time patients had access to that type of product was gel "A", "B" or "C". The evaluator of DH in no time knew what the gel ("A", "B" or "C") each patient was using. For this, the investigators asked the patients and the evaluator not talked about which product code they were using. In order to maintain blinding, randomization, control of compliance and verification of possible adverse reactions was performed by another reviewer (R.A.).

EXPERIMENTAL PROCEDURES

At Baseline, all patients received a supragingival prophylaxis with a rubber cup (Microdont®, São Paulo , SP , Brazil) and prophylactic paste (Villevie® , Joinville , SC , Brazil) . The products tested were always delivered in a transparent plastic syringe with 10 mls marking identified by the letters "A" , " B " or " C " . The syringes were given to individuals in an opaque plastic envelope sealed and delivered along with a reminder of the correct way to use the products. Guidance for the use of substances was to make application with a new toothbrush, 1 time a day (at night, before bed, after brushing the teeth) with the product received, for 1 minute and the amount of 0.25 g (0.5 ml) of the product as the demarcation the syringe. It was recommended that after using the products, they were expelled without rinsing the oral cavity with water.

All the dependet variables (Primary and secundary) were evaluated at baseline, 7, 15 and 30 days. A week before the baseline study, a dentifrice (Colgate Triple Action, Colgate - Palmolive , São Paulo , Brazil; 1450 ppm fluoride, abrasives: calcium carbonate , sodium bicarbonate and sodium silicate) was made available to all patients. This wash-out period was adopted to minimize interference from any other product with specific action to DH during the trial period. At baseline, was made available to all participants a new soft-bristled toothbrush, tufts in one direction and bristles rounded finish (professional Colgate Extra Clean , Colgate - Palmolive , São Paulo , Brazil). It was recommended that oral hygiene was performed three times a day just with toothbrush, toothpaste and floss without the use of mouthwashes. They recommended the use of 0.5 grams of toothpaste on the brush (Fill in the horizontal width of the brush with toothpaste).

Survey participants were instructed to return to the reviews of 7, 15 and 30 days bringing their new toothbrush, so was performed plaque removal site before testing the DH.

COMPLIANCE CONTROL

It was initially demonstrated by examining the amount of product to be used with an empty syringe. Adherence to treatment was performed with the control of the use of the substance by the inner end of the syringe plunger. In each evaluation, the patient returned with a syringe containing part of the product. In 7-day trial syringe should be rolled 6.5 ml, 2.5 ml at 15 days (in this assessment the patient received another syringe containing 5ml of the product), and at 30 days the two syringes should be empty. To maintain blinding of the examiner, the control of adherence was performed by the same person who made the randomization (R.A.).

DATA ANALYSIS

The unit of analysis was the individual. Means and 95% confidence intervals of the VASs in different stimuli were described for each group and experimental time. It was also verified the reduction of DH by subtracting the VAS of day 30 for the baseline VAS (delta) for each experimental group. After the data normality test, nonparametric tests were applied. Mean VASs of each experimental group were compared using the Kruskal-Wallis and Mann-Whitney test. Within-group analyzes at different time points were compared using the Wilcoxon test. Still, the VAS was dichotomized to "Take Pain" (VAS ≤ 25) and "Moderate pain / severe" (VAS> 25) and intergroup comparisons were performed using chi-square test. The level of significance was set at 5%. Data were analyzed by statistical software PASW Statistics Data Editor 17.0 (Statistical Package for the Social Sciences, PASW, Chicago, Ill).

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals who had been considered with a tooth with gingival recession and DH caused by at least one of the stimuli, heat (air), tactile (probe) and/or osmotic (water). If the subject submit more than one tooth with DH, the most sensitive element to the air test was chosen as the unit of analysis. Molars were excluded from analysis.

Exclusion Criteria:

* Ineligible individuals were characterized by exhibiting one of the following conditions:
* Had undergone periodontal surgery in the last three months;
* Chronic use of anti-inflammatory and analgesic,
* Receiving specific treatment for DH,
* Presented hypersensitivity to any of the compounds used in the study;
* Pregnant or lactating;
* Systemic conditions that could cause or predispose the development of DH (oesophageal reflux);
* subjects whose diet submit excess acidic substances;
* Persons whose tooth with DH present carie cavities, fractures, pulp necrosis or some pulp symptoms diagnosed through pulp sensitivity tests to cold;
* Present congenital defects in enamel or dentin;
* Present extensive restoration carried out in the last three months
* Present dental crowns and abutment of fixed or removable prosthesis.

Exclusion criteria after the start of the study:

* Patients who did not returned calls for the achievement of sensitivity tests in the stipulated period;
* Individuals that did not use adequadely the product;
* Subjects that desist from participating in the search, for any reason.
* Participants who presented worsening of DH;
* Subjects that presented some kind of reaction was observed, irritation or allergy to any of the products.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
dentine hypersensitivity with visual analog scale (VAS) following tactile, thermal and osmotic stimulus | Change from Baseline in VAS Scale at 7 days.
  The DH was measured on 7 days after products use. It was evaluated on the buccal surface of the tooth selected using a visual analog scale (VAS) immediately after application of the air jet, created with the triple syringe, at a distance of 10 mm from the tooth for 10 seconds, in the region of exposure root. The touch test was performed on the exposed root surface by applying a light force with blunt probe perpendicular to the long axis of the tooth for 10 seconds. Finally, we applied the test with water jet, using the perpendicular triple syringe and spaced 10 mm of the tooth to be tested. DH evaluations were performed with an interval of 1 minute to minimize interactions between examinations. All reviews of DH were conducted by a single trained examiner (M.M.).
dentine hypersensitivity with visual analog scale (VAS) following tactile, thermal and osmotic stimulus | Change from Baseline in VAS Scale at 15 days.
  he DH was measured on 15 days after products use. It was evaluated on the buccal surface of the tooth selected using a visual analog scale (VAS) immediately after application of the air jet, created with the triple syringe, at a distance of 10 mm from the tooth for 10 seconds, in the region of exposure root. The touch test was performed on the exposed root surface by applying a light force with blunt probe perpendicular to the long axis of the tooth for 10 seconds. Finally, we applied the test with water jet, using the perpendicular triple syringe and spaced 10 mm of the tooth to be tested. DH evaluations were performed with an interval of 1 minute to minimize interactions between examinations. All reviews of DH were conducted by a single trained examiner (M.M.).
dentine hypersensitivity with visual analog scale (VAS) following tactile, thermal and osmotic stimulus | Change from Baseline in VAS Scale at 30 days.
  The DH was measured on 30 days after products use. It was evaluated on the buccal surface of the tooth selected using a visual analog scale (VAS) immediately after application of the air jet, created with the triple syringe, at a distance of 10 mm from the tooth for 10 seconds, in the region of exposure root. The touch test was performed on the exposed root surface by applying a light force with blunt probe perpendicular to the long axis of the tooth for 10 seconds. Finally, we applied the test with water jet, using the perpendicular triple syringe and spaced 10 mm of the tooth to be tested. DH evaluations were performed with an interval of 1 minute to minimize interactions between examinations. All reviews of DH were conducted by a single trained examiner (M.M.).

SECONDARY OUTCOMES:
Irritation | Change from Baseline in possible adverse reactions at 7 days.
  Irritation was measures by interview and by clinical exam.
Irritation | Change from Baseline in possible adverse reactions at 15 days.
  Irritation was measures by interview and by clinical exam.
Irritation | Change from Baseline in possible adverse reactions at 30 days.
  Irritation was measures by interview and by clinical exam.
Allergy | Change from Baseline in possible adverse reactions at 07 days.
  Irritation was measures by interview and by clinical exam.
Allergy | Change from Baseline in possible adverse reactions at 15 days.
  Irritation was measures by interview and by clinical exam.
Allergy | Change from Baseline in possible adverse reactions at 30 days.
  Irritation was measures by interview and by clinical exam.
Bad taste | Change from Baseline in possible adverse reactions at 07 days.
  Irritation was measures by interview.
Bad taste | Change from Baseline in possible adverse reactions at 30 days.
  Irritation was measures by interview.

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio B Zanatta, pHD, Study Director — Universidade Federal de Santa Maria; ALESSANDRA P GRELLMANN, DS, Study Chair — Universidade Federal de Santa Maria; ROBERTO C VIANNA SANTOS, pHD, Study Chair — Centro Universitário Franciscano
Locations (1):
- Fabricio Batistin Zanatta, Santa Maria, Rua Floriano Peixoto--, Brazil